CLINICAL TRIAL: NCT05882149
Title: Randomized, Double-blind, Parallel, Placebo-controlled Study to Evaluate the Efficacy of Single Strain Probiotic, Delivered in a Chewing Gum, on the Reduction of Anthropometric Adiposity Biomarkers and the Improvement of Glucose Homeostasis in Abdominally Obese Individuals.
Brief Title: Single Strain Probiotic
Acronym: CHOICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rosa Sola (Other)
Collaborators: Biopolis S.L. (Industry); Chic-kles Gum, S.L. (Industry)
Responsible Party: Sponsor-Investigator, Rosa Sola, Doctor, full professor, University Rovira i Virgili
Organization: University Rovira i Virgili (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 074/2023
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-06

CONDITIONS: Abdominal Obesity
Keywords: waist circumference; visceral fat; probiotic supplementation; chewing gum
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel, placebo-controlled intervention study. The total duration of the intervention will be 12 weeks. The study will have two arms of intervention.
  The intervention product will be: sugar-free chewing gum with single strain probiotic and zinc.
  The Placebo product will be: sugar-free chewing gum. The placebo products and the intervention products will present the same format and appearance, in order to ensure the double-blind intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Sugar-free chewing gum with single strain probiotic and zinc. A daily dose of 2 chewing gums containing 1x10^10 Colony Forming Unit (CFU) for 12 weeks.
  Interventions: Dietary Supplement: Single strain probiotic
- Placebo (Placebo Comparator): Sugar-free chewing gum for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Single strain probiotic — Sugar-free chewing gum with single strain probiotic and zinc.
  The dosage will be 2 chewing a day, served at the same time and chewed for 6 minutes outside meals (for example 2h after breakfast or lunch).
  Arms: Probiotic
Dietary Supplement: Placebo — Sugar-free chewing gum.
  The dosage will be 2 chewing a day, served at the same time and chewed for 6 minutes outside meals (for example 2h after breakfast or lunch).
  Arms: Placebo

SUMMARY:
Probiotics have been recognized as functional foods with beneficial effects against obesity and cardiometabolic diseases, such as dyslipidemia, type 2 diabetes and the reduction of visceral fat mass, body weight and waist circumference.

In previous studies, it was shown that capsule/powder probiotic or postbiotic supplementation containing a single strain probiotic, could reduce anthropometric parameters, including the visceral fat area, and contribute to type 2 diabetes management in subjects with abdominal obesity. Similar findings were found when this single strain probiotic was delivered through enriched seafood sticks. Results showed that enriched seafood sticks significantly reduced insulin concentrations and HOMA-IR, pulse pressure, waist circumference, body weight and triglycerides.

These findings suggest that this specific single strain probiotic as a probiotic or postbiotic, could be a complementary strategy in the management of cardiometabolic disease risk factors.

Probiotics have mostly been studied incorporated in dairy food matrix. Other food matrices, such as chewing gum, have scarcely been exploited by the food industry. Chewing gum as a novel vehicle for probiotics presents the ability to release active ingredients into the oral cavity with a steady and rapid action. Furthermore, it has a high acceptance amongst adults and children and present few side effects.

No previous randomized controlled trials have examined the effect of a probiotic chewing gum on anthropometric adiposity biomarkers and glucose homeostasis in abdominally obese individuals.

The main objective of the present study is to evaluate the efficacy of single strain probiotic in the reduction of waist circumference in abdominally obese individuals.

The specific objectives:

* To evaluate the efficacy of single strain probiotic in the improvement of other anthropometric biomarkers (waist-hip-ratio, body weight, BMI, total fat mass, visceral fat index, free fat mass, lean body mass, conicity index, visceral adipose tissue and subcutaneous fat).
* To evaluate the efficacy of single strain probiotic in the management of glucose homeostasis.
* To evaluate the efficacy of single strain probiotic in the management of serum lipid levels.
* To evaluate the efficacy of single strain probiotic in the reduction of blood pressure and pulse pressure.
* To asses Quality of life after single strain probiotic supplementation.
* To identify changes in caloric intake and subjective satiety after single strain probiotic supplementation.
* To identify changes in gastrointestinal health after single strain probiotic supplementation.
* To identify changes in the oral microbiome after single strain probiotic supplementation.
* To identify changes in the gastrointestinal microbiome after single strain probiotic supplementation.

DETAILED DESCRIPTION:
A total of 180 adult volunteers will be included in the intervention (90 in each arm of the intervention).

During the CHOICE study, there will be 6 visits in total. Of these visits, 3 will be face-to-face and 3 by telephone. The study visits will be the following: screening visit (V0, face-to-face): to check inclusion/exclusion criteria and, in case of satisfying the inclusion criteria; basal visit (V1, face-to- face); visits during the intervention (V2, V3 and V4 via telephone); final study visit (V5, face-to-face).

In visits V0, V1 and V5 volunteers must present themselves in fasting conditions of 8 hours to obtain blood samples. In visits V1 and V5 volunteers must bring saliva and faeces samples.

In order to measure the changes in visceral adipose tissue, up to five days prior to the visit V1 and approximately up to 3 days prior after the V5, volunteers must have a Nuclear Magnetic Resonance (NMR) for measuring visceral fat.

CHOICE Study

Visit 0 (V0, week -1): Recruitment and selection

* Information to the volunteer and signature of the informed consent.
* Revision of the inclusion/exclusion criteria.
* Elaboration of study clinical history.
* Vital signs (blood pressure/resting heart rate).
* Checking the concomitant medication.
* Anthropometry (waist circumference; hip; body weight and composition; height).
* Blood sample extraction.
* Delivery of the 3-day dietary record and the material for feaces and saliva sample recollection for V1.
* Schedule the first visit and instructions (fasting).

Visit 1 (V1, week 0): Basal visit

* NMR (±5 days V1).
* Revision of study clinical history.
* Vital signs (blood pressure/resting heart rate).
* Checking the concomitant medication.
* Anthropometry (waist circumference; hip; body weight and composition).
* Blood sample extraction.
* Abdominal fat Ultrasound.
* Checking the 3-day dietary record.
* Checking the Three Factor Eating Questionnaire (TFEQ).
* Checking the Bing Eating Scale (BES).
* Checking the satiety scale (VAS) and gastrointestinal health information.
* Collection of feaces samples.
* Collection of saliva samples.
* Delivery of the 3-day dietary record and the material for saliva and feaces sample for V5.
* Schedule the next telephone visit and also the final visit and instructions (fasting).

Visit 2 (V2, week 3): Follow-up during the intervention

* Checking the concomitant medication.
* Record adverse effects.
* Checking adherence to product consumption (treatment compliance)
* Checking the satiety scale.
* Checking the gastrointestinal health.
* Schedule the next visit and instructions.

Visit 3 (V3, week 6): Follow-up during the intervention

* Checking the concomitant medication.
* Record adverse effects.
* Checking adherence to product consumption (treatment compliance)
* Checking the satiety scale.
* Checking the gastrointestinal health.
* Schedule the next visit and instructions.

Visit 4 (V4, week 9): Follow-up during the intervention

* Checking the concomitant medication.
* Record adverse effects.
* Checking adherence to product consumption (treatment compliance)
* Checking the satiety scale.
* Checking the gastrointestinal health.
* Schedule the next visit and instructions (fasting).

Visit 5 (V2, week 12): Final visit

* NMR (±3 days before V5).
* Revision of study clinical history.
* Vital signs (blood pressure/resting heart rate).
* Anthropometry (waist circumference; hip; body weight and composition)
* Checking the concomitant medication.
* Blood sample extraction.
* Abdominal fat Ultrasound.
* Checking the 3-day dietary record.
* Checking the TFEQ.
* Checking the BES.
* Record of adverse effects.
* Checking the treatment compliance
* Checking the satiety scale. (VAS)
* Collection of feaces samples.
* Collection of saliva samples.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 18 years old.
2. Established diagnosis of abdominal obesity: waist circumference (WC) ≥ 102 cm for men and ≥ 88 cm for women.
3. Voluntary, written, signed, informed consent to participate in the study.
4. Agreement to comply with the protocol and study restrictions.
5. Females of child-bearing potential require to provide a negative urine pregnancy test.

Exclusion Criteria:

1. WC < 102 cm for men, <88 cm for women, and >150 cm.
2. BMI ≥ 40 kg/m2.
3. Diagnosed and pharmacologically-treated type 1 or type 2 diabetes (fasting blood glucose ≥ 7 mmol/l).
4. Subjects with serious autoimmune disease, cardiovascular disease, liver dysfunction/disease, kidney dysfunction/disease, dementia, pancreatic disease, history of cancer within past 5 years, anemia, or any other disease or condition which, in the Investigator's opinion, could interfere with the results of the study or the safety of the subject.
5. Immunosuppression or ongoing therapy causing immunosuppression.
6. Pharmacologically-treated (medication/supplements) dyslipidemia.
7. Subjects consuming antibiotics in the previous 1 month.
8. Subjects consuming probiotics and prebiotics at least 1 month prior to inclusion in the study or during the intervention period.
9. Use of drugs or supplements to manage body weight or body fat in the last 3 months.
10. Use of laxatives or fiber supplements in the past 4 weeks.
11. History of chronic active inflammatory disorders.
12. History of bariatric surgery.
13. History of any chronic gastrointestinal disease (e.g. IBD).
14. Regular use of systemic or inhaled corticosteroids, or systemic immunomodulatory drugs.
15. Significant change in tobacco, snuff, nicotine and e-cigarette use habits in the past 3 months or planned cessation of the use of these products during the trial.
16. Active or recent (last 3 months) participation in a weight loss program (diet and/or exercise).
17. Weight change (increase or loss) of 3 kg during the past 3 months.
18. Pregnant or planning pregnancy during the study or breastfeeding.
19. Participation in a clinical trial with an investigational product or drug within 60 days prior to screening.
20. Illicit drug users.
21. Alcohol abusers.
22. Known hypersensitivity to any ingredients in the active or placebo products.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in waist circumference | From week 0 to Week 12
  Difference in waist circumference (cm) measured at the umbilicus using a 150-cm anthropometric steel measuring tape from week 0 to week 12

SECONDARY OUTCOMES:
Change in hip circumference | From week 0 to Week 12
  Differences in hip circumference (cm) measured at the widest portion of the buttocks using a 150-cm anthropometric steel measuring tape from week 0 to week 12
Change in waist-hip-ratio | From week 0 to Week 12
  Differences in waist-hip-ratio (cm) measured as waist circumference/hip circumference from week 0 to week 12
Change in Body weight | From week 0 to Week 12
  Differences in body weight (kg) measured using a Tanita MC 780-MA; Tanita Corp., Barcelona, Spain, from week 0 to week 12
Change in Body mass index | From week 0 to Week 12
  Differences in body mass index (kg/m2) calculated as weight (kg) divided to height (m2), from week 0 to week 12
Change in Total fat mass | From week 0 to Week 12
  Differences in total fat mass (% kg) measured using a Tanita MC 780-MA; Tanita Corp., Barcelona, Spain, from week 0 to week 12
Change in Free fat mass | From week 0 to Week 12
  Differences in free fat mass (%, kg) measured using a Tanita MC 780-MA; Tanita Corp., Barcelona, Spain, from week 0 to week 12
Change in Lean body mass | From week 0 to Week 12
  Differences in Lean body mass (%, kg) measured using a Tanita MC 780-MA; Tanita Corp., Barcelona, Spain, from week 0 to week 12
Change in Visceral fat index | From week 0 to Week 12
  Differences in visceral fat index obtained using a Tanita MC 780-MA; Tanita Corp., Barcelona, Spain, from week 0 to week 12
Change in Conicity index | From week 0 to Week 12
  Differences in Conicity index calculated as waist circumference (cm)/0.109 x square root of weight (kg)/height (m) from week 0 to week 12
Change in Visceral adipose tissue | From week 0 to Week 12
  Differences in Visceral adipose tissue (cm2) measured by MRI (transverse body scan in one axial slice 5cm over L5-S1) from week 0 to week 12
Change in Subcutaneous fat | From week 0 to Week 12
  Differences in Subcutaneous fat (cm2) measured by MRI, transverse body scan in one axial slice 5cm over L5-S1 from week 0 to week 12
Changes in Fasting blood glucose | From week 0 to Week 12
  Differences in Fasting blood glucose (mmol/L) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in Fasting insulin | From week 0 to Week 12
  Differences in Fasting insulin (IU/mL) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in HOMA index | From week 0 to Week 12
  Differences in HOMA index measured with the formula insulin x glucose/405 from week 0 to week 12
Changes in glycosylated hemoglobin (HbA1c) | From week 0 to Week 12
  Differences in glycosylated hemoglobin (%) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in Total cholesterol | From week 0 to Week 12
  Differences in Total cholesterol (mmol/L) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in HDLc | From week 0 to Week 12
  Differences in HDLc (mmol/L) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in LDLc | From week 0 to Week 12
  Differences in LDLc (mmol/L) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in Total Triglycerides | From week 0 to Week 12
  Differences inTotal Triglycerides (mmol/L) measured by Standardized methods in an automated analyzer from week 0 to week 12
Changes in Systolic blood pressure | From week 0 to Week 12
  Differences in Systolic blood pressure (mmHg) measured by an automatic phygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain) measured twice after adult respite 2-5 min seated, with a 1-min interval in between from week 0 to week 12
Changes in Diastolic blood pressure | From week 0 to Week 12
  Differences in Diastolic blood pressure (mmHg) measured by an automatic hygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain) measured twice after adult respite 2-5 min seated, with a 1-min interval in between from week 0 to week 12
Changes in Pulse Pressure | From week 0 to Week 12
  Differences in Pulse pressure (mmHg), calculated as the difference between the upper and lower numbers of blood pressure, from week 0 to week 12
Changes in Three Factor Eating Questionnaire (TFEQ; Spanish edition) | From week 0 to Week 12
  Differences in TFEQ score from week 0 to week 12. The minimum score is 0 and maximum score is 100, and higher score means a worse outcome.
Changes in Bing Eating Scale (BES; Spanish edition) | From week 0 to Week 12
  Differences in BES score from week 0 to week 12. The minimum score is 0 and maximum score is 46, and higher score means a worse outcome.maximum score is 100, and higher score means a worse outcome.
Changes in dietary intake | From week 0 to week 12
  Differences in dietary intake assessed by a 3-day dietary record from week 0 to week 12
Changes in Satiety | From week 0 to week 3, week 6, week 9 and week 12
  Differences in satiety, assessed by a Visual Annual Scale (VAS), from week 0 to week 3, week 6, week 9 and week 12. The minimum score is -100 mm and maximum score is 100 mm, and higher score means a better outcome.
Changes in bowel habit | From week 0 to week 3, week 6, week 9 and week 12
  Differences in bowel habit, assessed by bristol scale, from week 0 to week 3, week 6, week 9 and week 12. In this scale there are 7 descriptive points, the minimum score is "severe constipation" and maximum score is "severe diarrhea". The better outcome is in the middle of the 7 descriptive points (points 3 and 4): "normal".
Changes in flatulences | From week 0 to week 3, week 6, week 9 and week 12
  Differences in the presence of flatulence (yes or not), from week 0 to week 3, week 6, week 9 and week 12
Changes in nausea | From week 0 to week 3, week 6, week 9 and week 12
  Differences in the presence of nausea (yes or not), from week 0 to week 3, week 6, week 9 and week 12
Changes in reflux | From week 0 to week 3, week 6, week 9 and week 12
  Differences in the presence of reflux (yes or not), from week 0 to week 3, week 6, week 9 and week 12
Changes in abdominal distension | From week 0 to week 3, week 6, week 9 and week 12
  Differences in the presence of abdominal distension (yes or not), from week 0 to week 3, week 6, week 9 and week 12
Changes in diarrhea | From week 0 to week 3, week 6, week 9 and week 12
  Differences in the presence of diarrhea (yes or not), from week 0 to week 3, week 6, week 9 and week 12
Changes in gut microbiota | From week 0 to week 12
  Differences in Phyla composition, assessed by metagenomics, from week 0 to week 12
Changes in oral microbiota | From week 0 to week 12
  Differences in Phyla composition, assessed by metagenomics, from week 0 to week 12
Change in Visceral adipose tissue | From week 0 to week 12
  Differences in Visceral adipose tissue (mm) measured by ultrasound (xipho-umbilical axis, 1-5 cm above navel) from week 0 to week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Ten Hoevel C, Besora-Moreno M, Queral J, Llaurado E, Valls RM, Sola R, Pedret A. Ultrasound and MRI abdominal fat distribution and its associations with metabolic conditions in adults with abdominal obesity. Diabetes Obes Metab. 2025 Dec 17. doi: 10.1111/dom.70390. Online ahead of print. PMID 41403258